CLINICAL TRIAL: NCT01619488
Title: Laparoscopic Adjustable Gastric Banding for Treatment of Morbid Obesity in Adolescents
Brief Title: Laparoscopic Adjustable Gastric Banding in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirk Reichard (Other)
Responsible Party: Sponsor-Investigator, Kirk Reichard, OR SURGICAL DIRECTOR, Nemours Children's Clinic
Organization: Nemours Children's Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0082295
Record Dates: First submitted 2012-06-07; First posted 2012-06-14 (Estimated); Results first posted 2023-06-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Morbid Obesity
Keywords: Lap-Band; morbid obesity; adolescents
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gastric Banding (Experimental): Surgical placement of an adjustable gastric band around the upper portion of the stomach.
  Adjustments are made to the band through a subcutaneous port as needed to maintain appropriate restriction.
  Interventions: Device: Adjustable Gastric Band

INTERVENTIONS:
Device: Adjustable Gastric Band — Surgical placement of an adjustable gastric band around the upper portion of the stomach.
  Adjustments are made to the band through a subcutaneous port as needed to maintain appropriate restriction.
  Other Names: Lap-Band

SUMMARY:
This study is to determine if the Lap-band system is safe and effective for use in morbidly obese adolescents.

DETAILED DESCRIPTION:
This study is to determine if the Lap-band system is safe and effective for use in morbidly obese adolescents

ELIGIBILITY:
Inclusion Criteria:

* ages 14-19
* BMI > 35
* history of obesity for at least 5 years with failed attempts at diet and medical management for at least 6 months.
* confirmation by a pediatric psychologist that the subject is sufficiently mature emotionally and has adequate family support to comply with the study protocol.

Exclusion Criteria:

* history of congenital or acquired anomalies of the GI tract.
* history of esophageal motility disorders
* uncontrolled psychiatric problems
* previous esophageal, gastric or bariatric surgery; intestinal obstruction or peritonitis.
* uncontrolled eating disorders

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2007-04-23 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Reichard, MD, Principal Investigator — A I duPont Hospital for Children; Nemours Children's Clinic
Locations (1):
- A I duPont Hospital for Children/Nemours Children's Clinic, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were recruited from the pediatric weight management clinic.
Pre-assignment Details: Of 136 eligible patients, 57 completed the pre-intervention program and underwent placement of the gastric band. The remainder opted out of the intervention.
Groups:
- Gastric Banding: Surgical placement of an adjustable gastric band around the upper portion of the stomach.
  Adjustments are made to the band through a subcutaneous port as needed to maintain appropriate restriction.
  Adjustable Gastric Band: Surgical placement of an adjustable gastric band around the upper portion of the stomach.
  Adjustments are made to the band through a subcutaneous port as needed to maintain appropriate restriction.
Period: Overall Study
Arm/Group | Gastric Banding
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gastric Band: Lap Band Surgery was ultimately performed on 57 patients, the remainder chose alternative management.
Arm/Group | Gastric Band
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.05 (1.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 37
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 57
Weight [Mean (Standard Deviation); unit: Kilogram] | 139.36 (19.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Weight Loss
Description: Weight loss in kilograms Weight on day of surgery minus last weight recorded before end of trial
Time Frame: Up to five years post surgery.
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Weight Loss: 57 Patients who underwent Adjustable gastric band surgery
Arm/Group | Weight Loss
Number analyzed (Participants) | 57
kilograms | 11.35 (19.08)

2. Secondary Outcome: Insulin Resistance
Description: Fasting insulin level
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: uIU/ml
Groups:
- Fasting Serum Insulin Change: Fasting serum insulin obtained at study entry minus level at 12 month visit
Arm/Group | Fasting Serum Insulin Change
Number analyzed (Participants) | 57
uIU/ml | 12.5 (14.0)

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Adverse Events: 2 Adverse events requiring successful removal of band for slipped bands.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 2/57
Other Adverse Events (participants affected / at risk) | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=57)
Band slippage, leading to removal (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes